CLINICAL TRIAL: NCT03544606
Title: Nitric Oxide Donor Isosorbide Mono Nitrate for Cervical Ripening in Induction of Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ahmed nagy shaker ramadan (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Sponsor-Investigator, ahmed nagy shaker ramadan, director, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ISMN and labor induction
Record Dates: First submitted 2018-05-18; First posted 2018-06-04 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — isosorbide-5-mononitrate; Pyridoxine

STUDY DESIGN:
Intervention Model Description: The patients will be divided into 2 groups.
  Group 1:
  80 pregnant females, induction of labor will be done by Intra vaginal isosorbide mono nitrate (Effox 40 mg MINAPHARM)
  Group 2:
  80 pregnant females, induction will be done by placebo (pyridoxine) administered in the posterior vaginal fornix.
Who Masked: Participant, Care Provider
Masking Description: To insure that everyone has the chance of participation, Randomization will be done using computer generated randomization sheet using statsdirect version 3. Double blinding will be done by one of the supervisors who will be the only one to know the key, thus the care provider and the patient will not know is it the drug or the placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isosorbide mononitrate group (Experimental): In vaginal IMN group (group 1) 40 mg tablet of intra-vaginal IMN (Effox; MINAPHARMA, Cairo, Egypt) will be placed into the posterior fornix of the vagina, through a digital vaginal examination, every 4 h for a maximum of four doses.
  Interventions: Drug: isosorbide mononitrate
- placebos group (Placebo Comparator): In the placebo group (group 2) 40 mg intra-vaginal pyridoxine placebos every 4 h for a maximum of four doses will be given
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: isosorbide mononitrate — 40 mg tablet of intra-vaginal IMN (Effox; MINAPHARMA, Cairo, Egypt) will be placed into the posterior fornix of the vagina, through a digital vaginal examination, every 4 h for a maximum of four doses.
  Other Names: Effox 40 mg
  Arms: isosorbide mononitrate group
Drug: Placebos — In placebo group (group 2) 40 mg intra-vaginal pyridoxine placebos every 4 h for a maximum of four doses will be given
  Other Names: pyridoxine
  Arms: placebos group

SUMMARY:
The study aims to evaluate and assess the effectiveness and safety of vaginal administration of isosorbide mono nitrate (IMN) to induce cervical ripening and shorten the interval time between induction and delivery in women undergoing induction of labor.

Research Hypothesis:

In women undergoing induction of labor, vaginal administration of isosorbide mono nitrate (IMN) is effective to induce cervical ripening and shorten the interval time between induction and delivery.

Research Questions:

Does vaginal administration of isosorbide mono nitrate (IMN) induce cervical ripening and shorten the interval time between induction and delivery in women undergoing induction of labor?

DETAILED DESCRIPTION:
* Type of Study : Prospective double blind randomized controlled clinical trial.
* Study Setting : This study will be conducted in Kafr Elsheikh University maternity hospital.
* Study Period : Expected 6 months from December 2023 to June 2024.
* Study Population : Patients will be recruited in this study those attending labor ward at Kafr Elsheikh hospital for induction of labor at term or post-term with unripe cervix (Bishop Score ˂ 6).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Cephalic presentation.
* Bishop score < 6.
* Average size of the fetus.
* Adequate pelvic dimensions.
* Term or post-term pregnancies with an indication for labor induction either maternal or fetal.

Exclusion Criteria:

* • Previous uterine scar.

  * Patients with regular uterine contractions.
  * Malpresentation.
  * Multifetal gestation.
  * Prelabour rupture of membranes.
  * Established fetal distress.
  * Indication for CS, e.g. Major degree of cephalopelvic disproportion and fetal macrosomia.
  * Antepartum hemorrhage.
  * Active genital herpes infection.
  * Severe maternal illness (e.g. severe preeclampsia).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
admission-delivery interval | up to 24 hours
  The time from initiation labor induction and delivery of placenta

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed N Shaker, MD, Principal Investigator — faculty of medicine - Kafr elsheikh university
Locations (1):
- faculty of medicine - Kafr Elsheikh university, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
The data supporting this research is available upon request. Please contact corresponding Author at ahmedafifi38527@postgrad.kasralainy.edu.eg for access to the relevant datasets. We are committed to transparency and facilitating the reproducibility of our findings, and we welcome inquiries regarding the data used in this study.